CLINICAL TRIAL: NCT02427139
Title: Study of ANSiStim for Pain Relief During Active Labor Phase Through Continues Checking of VAS SCORE
Brief Title: ANSiStim Study for Active Labor Pain
Acronym: ANSS-ALP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: DyAnsys, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: ANSS-ALP 01
Record Dates: First submitted 2015-04-21; First posted 2015-04-27 (Estimated); Last update posted 2016-05-24 (Estimated); Status verified 2016-05

CONDITIONS: Labor Pain; Obstetric Pain
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ANSiStim (Experimental): The ANSiStim device is designed to administer auricular point stimulation treatment over several days. The advantage of using the ear for this treatment is that it provides numerous points for stimulation within a small area. Stimulation is performed by electrical pulses emitted through strategically positioned needles.
  Three zinc air batteries with 1.4 V provide the required stimulation energy for 96 hours. This constant current source guarantees equivalent stimulation energy regardless of the individual impedance of the skin. The treatment period varies based on the severity of the pain. To minimize the risk of adaption or tolerance to the electrical stimulation, it is applied for 3 hours, followed by a pause of 3 hours.
  Interventions: Device: ANSiStim

INTERVENTIONS:
Device: ANSiStim — ANSiStim allows continuous point stimulation over a period of several days while offering the patient a high degree of comfort and mobility at the same time. Use of the ANSiSTIM therapy provides overwhelming advantage over drug therapy minimizing possible side-effects caused by pain medications (i.e. opioid) such as, for example, impaired reactions. In most cases, the patient continues to lead its life as normal, without side effects or any loss of quality of life.

SUMMARY:
The specific aim of the study is to do comparison between ANSiStim and Placebo for pain relief in labor. During the treatment, pain relief will be assesed with ANSiStim in active labor through continues checking of VAS SCORE. ANSiStim has been tried in post operative patients with good pain relief .

DETAILED DESCRIPTION:
Pain during labor is caused by contractions of the muscles of the uterus and by pressure on the cervix. This pain can be felt as strong cramping in the abdomen, groin, and back, as well as an achy feeling. Some women experience pain in their sides or thighs as well. Most women have an epidural or spinal during labour or after the birth.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant Women on an Active Labor

Exclusion Criteria:

* Cardiac Pacemaker or any other implants
* Psoriasis
* Diminish mental capacity

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Evidence of Reduced Pain (Pain Scale of 5) in Active Labor Phase after ANSiStim Placement | 48 Hours

CONTACTS AND LOCATIONS:
Overall Officials: Gayathri D Kamath, M.D., Principal Investigator — Fortis Hospital - Bangalore
Locations (1):
- Fortis Hospital, Bangalore, Karnataka, India